CLINICAL TRIAL: NCT04179929
Title: Treatment of BCR-ABL Negative ALL in Adults According to MRD and Genetics
Brief Title: Treatment of Breakpoint Cluster Region-Abelson (BCR-ABL) Negative ALL in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA LAL-2019
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; adult; Ph-negative; minimal residual disease; transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHEMOTHERAPY (Other): Pediatric-type of chemotherapy
  Interventions: Drug: Pediatric-type of chemotherapy
- allogeneic HSCT (Other): allogeneic HSCT
  Interventions: Procedure: allogeneic HSCT

INTERVENTIONS:
Drug: Pediatric-type of chemotherapy — Pediatric type chemotherapy (induction, early and delayed consolidation, reinduction, maintenance). Induction (VCR,PDN,PegASP,DNR). Early and delayed consolidation (high-dose Methotrexate, high-dose Cytarabine, PegASP). Reinduction (VCR, PDN, PegASP, DNR). Maintenance (Methotrexate, Mercaptopurine)
  Arms: CHEMOTHERAPY
Procedure: allogeneic HSCT — allogeneic HSCT
  Arms: allogeneic HSCT

SUMMARY:
After consolidation therapy adult patients (≥18 yr) with Ph-negative ALL will be treated with continuation chemotherapy or allogeneic hematopoietic stem cell transplantation (alloHSCT) according to both measurable residual disease (MRD) and results of genetic study performed at baseline.

DETAILED DESCRIPTION:
Patients will be uniformly treated with four drug-induction: vincristine (VCR), prednisone (PDN), pegylated asparaginase (PegASP), daunorubicin (DNR).

Resistant patients will receive a second induction with fludarabine, Ara-C, G-Colony-Stimulating Factor (G-CSF) and idarubicin (FLAG-IDA).

Patients with adequate MRD clearance after induction will receive 3 blocks of early consolidation. If adequate MRD clearance and good genetic background, the patients will proceed to delayed intensification, reinduction and maintenance. The remaining patients will receive early or delayed alloHSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-60 yr with de novo Ph-neg ALL
* Eastern Cooperative Oncology Group (ECOG) 0-2 (or >2 if due to ALL)
* Informed consent

Exclusion Criteria:

* Mature B-ALL, Ph+ ALL or blast crisis of chronic myeloid leukemia (CML), ALL of ambiguous lineage
* ECOG >2 not due to ALL
* Impaired cardiac, respiratory, hepatic or renal function not due to ALL
* Pregnancy
* HIV positivity
* Severe psychiatric disease
* Negative to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Time from diagnosis to death or last follow-up

SECONDARY OUTCOMES:
Complete remission (CR) rate | 4 or 8 weeks after treatment onset
  Proportion of patients who achieve CR with or 2 induction therapy lines
MRD status after induction and consolidation | After induction (4-8 weeks) and consolidation (16-20 weeks)
  Proportion of patients who achieve and maintain the negative MRD status (<10-4)

OTHER OUTCOMES:
alloSCT realization | Early alloHSCT: 15-20 weeks from diagnosis. Delayed: 30-35 weeks from diagnosis.
  Proportion of patients who receive early or delayed alloHSCT

CONTACTS AND LOCATIONS:
Locations (83):
- Spain (83):
  - Ico-Hugtip, Badalona, Barcelona
  - H. A Coruña, A Coruña
  - H Albacete, Albacete
  - H. General Univ. de Alicante, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Clínica Teknon, Barcelona
  - H del Mar, Barcelona
  - H. Clínic de Barcelona, Barcelona
  - H. del Mar, Barcelona
  - H. Sant Pau, Barcelona
  - H. Vall d'Hebron, Barcelona
  - ICO-Duran i Reynals, Bellvitge
  - H Basurto, Bilbao
  - Hu Basurto, Bilbao
  - H. Jerez, Cadiz
  - H. Puerta del Mar, Cadiz
  - H. General de Castellón, Castelló
  - H. San Pedro de Alcántara, Cáceres
  - H. Reina Sofía, Córdoba
  - H. Fuenlabrada, Fuenlabrada
  - H Galdakao, Galdakao
  - H. Univ. De Getafe, Getafe
  - ICO-Dr.Josep Trueta, Girona
  - H. Guadalajara, Guadalajara
  - H Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario Ciudad de Jaén, Jaén
  - H. Jerez de la Frontera, Jerez de la Frontera
  - H. General Lanzarote, Lanzarote
  - H Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hu Gran Canarias Dr Negrin, Las Palmas de Gran Canaria
  - H. Arnau De Vilanova, Lleida
  - H. Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - H La Zarzuela, Madrid
  - H Puerta de Hierro, Madrid
  - H. 12 de Octubre, Madrid
  - H. Clínico de Madrid, Madrid
  - H. Gregorio Marañón, Madrid
  - H. Infanta Sofía, Madrid
  - H. Madrid-Norte Sanchinarro, Madrid
  - H. Ramón y Cajal, Madrid
  - H. Univ La Paz, Madrid
  - Hu Infanta Leonor, Madrid
  - Hu La Princesa, Madrid
  - H. Carlos Haya, Málaga
  - H. Clínico Univ. Virgen de la Victoria, Málaga
  - H. Regional de Málaga, Málaga
  - H. Morales Meseguer, Murcia
  - H. Virgen de la Arrixaca, Murcia
  - Complejo Hosp. Univ. de Orense, Ourense
  - H. Central de Asturias, Oviedo
  - H Río Carrión, Palencia
  - H. Son Espases, Palma de Mallorca
  - H. Son Llàtzer, Palma de Mallorca
  - Complejo Hospitalario Navarra, Pamplona
  - H. Clínico Univ. de Navarra, Pamplona
  - H. Virgen del Camino, Pamplona
  - Complejo Hospitalario Pontevedra - Hospital Montecelo, Pontevedra
  - H. Parc Taulí, Sabadell
  - H. Clínico Univ. de Salamanca, Salamanca
  - H Donostia, San Sebastián
  - H. Univ. de Canarias, Santa Cruz de Tenerife
  - H. Marqués de Valdecilla, Santander
  - Complejo Hosp. Univ. Santiago de Compostela, Santiago de Compostela
  - H. General de Segovia, Segovia
  - H. Universitario de Valme, Seville
  - H. Virgen del Rocío, Seville
  - ICO-Joan XXIII, Tarragona
  - Mútua de Terrassa, Terrassa
  - H Torrejón, Torrejón de Ardoz
  - H. Verge de la Cinta, Tortosa
  - H. Arnau de Vilanova, Valencia
  - H. Clínico Univ. de Valencia, Valencia
  - H. Dr. Peset, Valencia
  - H. General Univ. de Valencia, Valencia
  - H. la Fe, Valencia
  - H. Clínico Universitario de Valladolid, Valladolid
  - H. Río Hortega, Valladolid
  - H. Xeral-Cíes Vigo, Vigo
  - H. Virgen de la Concha, Zamora
  - H. Lozano Blesa, Zaragoza
  - H. Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor of the study — https://www.fundacionpethema.es